CLINICAL TRIAL: NCT01449006
Title: A Randomised Controlled Clinical Trial of the Efficacy of HAART Intensification With Maraviroc in HIV Virally Suppressed Patients With Cognitive Impairment
Brief Title: A Study of the Neurological Effects of Adding Maraviroc to HAART Regimen in Patients With HIV (HANDmac)
Acronym: HANDmac
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bruce Brew (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Bruce Brew, Professor, St Vincent's Hospital
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/066; 114560 (Other Grant/Funding Number: VIIV Healthcare Australia)
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Associated Neurocognitive Disorders (HAND)
Keywords: HIV; HAND; Maraviroc; Neurocognitive; Neurology; Human Immunodeficiency Virus; HIV Associated Neurocognitive Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care HAART regimen (No Intervention): Participants randomised to this arm of the trial will remain on their usual prescribed HAART regimen.
- Maraviroc (Experimental): Participants randomised to this arm will remain on their usual prescribed HAART regimen, with the addition of Maraviroc. Maraviroc will be prescribed according to the Product Information Sheet, with consideration given to background therapy.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc oral tablet. Dosage: 150 mg twice daily, 300 mg twice daily, or 600 mg twice daily. Dosing will be dependent on the participant's background HAART therapy, and will be in accordance with the product information sheet.
  Other Names: Celsentri
  Arms: Maraviroc

SUMMARY:
HIV related cognitive impairment still occurs despite highly active antiretroviral therapy (HAART). HIV disease affects the brain in 20-40% of patients with advancing HIV disease; leading to varying degrees of cognitive impairment, recently termed HIV associated neurocognitive disorders (HAND). HAND may occur in patients who are virally suppressed in both blood and CSF.

Patients with HIV Associated Neurocognitive Disorders (HAND) who are virally suppressed in both their blood and cerebrospinal fluid (CSF), whilst on a highly active antiretroviral therapy (HAART) regimen may have significant cognitive improvement with HAART intensification with the medication Maraviroc; compared to those who remain on their existing regimen.

This study will be a prospective, interventional, randomised and unblinded controlled clinical trial. The aim of this study will be to determine whether HAART intensification with the medication Maraviroc, leads to significant improvement in HIV associated neurocognitive disorders (HAND).

Patients with the recent progression (within 6 months) of HAND (validated by neuropsychological assessment) on HAART, who are virally suppressed (<50 copies per ml) in blood and CSF will be randomised to have their existing HAART regimen intensified with Maraviroc, or not. The control arm will remain on their medication regimen as prescribed. The target is to enrol 70 patients into the control group, and 70 patients into the Maraviroc intensification group.

Patients will undergo baseline neuropsychological testing, MRI, blood tests, and cerebrospinal fluid (CSF) tests (via a lumbar puncture). The methods used to determine the effectiveness of adding Maraviroc, will include further neuropsychological assessment at 6 months, and neuropsychological assessment, MRI and CSF assessment again at 12 months.

Neuropsychological testing completed at 6 and 12 months will be completed by a "blind assessor", in that they will have no knowledge of which arm (treatment or control) the participant is enrolled in.

An evaluation (neuropsychological testing) will be performed should the patient deteriorate during the course of the study, as recognised by the patient's managing physician.

At the end of the study protocol (12 months) the patient's HAART therapy will be managed by their primary physician.

ELIGIBILITY:
Inclusion Criteria:

* HIV Positive
* On HAART, with plasma viral load < 50 copies/ml for previous 12 months or more
* Able to provide informed consent
* HAND diagnosis, with symptom progression within previous 6 months

Exclusion Criteria:

* Non-HIV related neurological disorders and active central nervous system (CNS) opportunistic infection (as assessed by full blood count, electrolytes, creatinine, glucose, liver funciton tests, cryptococcal antigen, venereal disease research laboratory (VDRL), MRI brain scan and CSF analysis for cell count, protein, glucose, culture, VDRL and cryptococcal antigen)
* Psychiatric disorders on the psychiatric axis
* Current major depression
* Current substance use disorder, or severe substance use disorder within 12 months of study entry
* Active Hepatitis C Virus (HCV) (detectable HCV RNA)
* History of loss of consciousness > 1 hour
* Non-proficient in English
* Medications known to pharmacologically interact with antiretrovirals (ARVs)
* Currently taking an entry inhibitor
* Pregnancy (as assessed by the urine pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Brew, MBBS, PhD, Principal Investigator — St Vincent's Hospital - Sydney, Australia
Locations (2):
- Australia (2):
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria

REFERENCES:
- [Result] Gates TM, Cysique LA, Siefried KJ, Chaganti J, Moffat KJ, Brew BJ. Maraviroc-intensified combined antiretroviral therapy improves cognition in virally suppressed HIV-associated neurocognitive disorder. AIDS. 2016 Feb 20;30(4):591-600. doi: 10.1097/QAD.0000000000000951. PMID 26825032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from St Vincent's Hospital and/or referred from tertiary sexual health centres over the period January 2012 to June 2013.
Pre-assignment Details: Two enrolled participants failed screening (1 HCV+, 1 not cognitively impaired)
Period: Overall Study
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Started | 8 | 9
Completed | 5 | 9
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data presented reflect baseline demographic and clinical characteristics for participants included in the primary analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care HAART Regimen | Maraviroc | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.4) | 52.2 (3.7) | 55 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 9 | 14
Education [Mean (Standard Deviation); unit: years] | 11.6 (2.3) | 12.3 (2.8) | 12.1 (2.6)
Premorbid intelligence quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — Full-scale IQ based on National Adult Reading Test (NART) error score. NART is a test of reading ability that has been extensively validated for use as a proxy measure of pre-morbid intellectual functioning. Full-Scale IQ score is expressed as a Standard Score with Mean=100 and Standard Deviation=15. Values range from 69-131. Higher scores indicate better performance.
  units on a scale | 104.4 (18.9) | 102.2 (16.3) | 103 (16.6)
Nadir cluster of differentiation 4 (CD4) [Median (Inter-Quartile Range); unit: cells/mm3] | 310 [51 to 390] | 150 [33.5 to 253.5] | 174.5 [36.8 to 312.5]
Current CD4 [Median (Inter-Quartile Range); unit: cells/mm3] | 980 [548 to 1041] | 499 [338 to 827.5] | 625.5 [400.8 to 979.3]
HAND Status [Number; unit: participants]
  Asymptomatic Neurocognitive Impairment (ANI) | 1 | 1 | 2
  Mild Neurocognitive Disorder (MND) | 2 | 8 | 10
  HIV-Associated Dementia (HAD) | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurocognitive Functioning
Description: Change in overall neurocognitive performance, defined as a global neurocognitive z-score, over the study time-period (baseline, 6-months, 12-months). To derive this score, 1) raw scores obtained from a 5-domain brief neurocognitive battery were converted to age-corrected z-scores (M=0, SD=1) and 2) the set of individual subtest z-scores were averaged to generate a single composite (global) z-score for each subject. Lower (negative) scores therefore indicate greater levels of cognitive impairment.
Time Frame: Baseline, 6-months and 12-months
Population: Modified intent-to-treat analysis. All randomized participants were included except for n=2 controls with baseline data only (1 lost to follow-up, 1 withdrew before 6-months) and n=1 control where a protocol violation was noted (randomized without conclusive evidence of neurocognitive impairment - see participant flow section).
Measure: Least Squares Mean (Standard Error); unit: Global Neurocognitive Z-Score
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Number analyzed (Participants) | 5 | 9
Global Neurocognitive Z-Score
  Baseline | -0.94 (0.30) | -0.81 (0.23)
  6 months | -1.03 (0.30) | -0.51 (0.23)
  12 months | -0.93 (0.30) | -0.56 (0.23)
Statistical Analysis 1: Comparison: Standard of Care HAART Regimen vs Maraviroc; The primary outcome was analysed using a mixed-effect regression model with arm and time as fixed linear effects, arm*time interaction as a non-linear fixed effect and participant as a random effect to account for participant attrition; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — This pilot study was conducted to generate effect sizes for a potential larger investigation. The study design and small sample size had limited power to detect a statistically significant effect at p<0.05, so no p-value threshold was strictly set; 41 data points included (control n=14; maraviroc: n=27); n=1 control did not attend 12-month visit
Statistical Analysis 2: Comparison: Standard of Care HAART Regimen vs Maraviroc; Clinical relevance of the effect size observed at 6-months was assessed by generating Cohen's d statistic and 90% confidence interval (CI) around the estimate; Test type: Superiority or Other; Cohen's d = 0.77, 90% CI 2-sided [-0.19 to 1.71] — Positive value reflects improved neurocognitive functioning in maraviroc arm compared to control arm
Statistical Analysis 3: Comparison: Standard of Care HAART Regimen vs Maraviroc; Clinical relevance of the effect size observed at 12-months was assessed by generating Cohen's d statistic and 90%CI around the estimate; Test type: Superiority or Other; Mean Difference (Final Values) = 0.55, 90% CI 2-sided [-0.47 to 1.55] — Positive value reflects improved neurocognitive functioning in maraviroc arm compared to control arm

2. Secondary Outcome: Change in CSF Neopterin Concentration
Description: Change in concentration of the CSF neuroinflammatory marker neopterin (measured in nmol/L) from baseline to 12-months.
Time Frame: Baseline and 12-months
Population: The analysis included all randomized participants who were included in the primary analysis aside from n=1 control and n=2 maraviroc who did not provide a CSF sample at 12-months.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Number analyzed (Participants) | 4 | 7
nmol/L
  Baseline | 11.5 (3.41) | 12.57 (2.57)
  12-months | 13.25 (3.41) | 15.71 (2.57)
Statistical Analysis 1: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in CSF neopterin levels was analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.82, ANOVA

3. Secondary Outcome: Change in MRS Cerebral Metabolite Ratios in Basal Ganglia
Description: Change in major cerebral metabolites in the basal ganglia, as measured by 1H-Magnetic Resonance Spectroscopy (MRS), between baseline and 12-months. Spectra were acquired on a Phillips Achieva 3T MRI scanner using point-resolved spectroscopy (PRESS) sequence with short echot time (TE). jMRUI/AMARES algorithm was used to process spectra. Metabolite ratios were calculated for the following metabolites: N-acetyl aspartate (NAA), choline (Cho), creatine (Cr), myo-inositol (mIo), in relation to internal water (H20) as standard.
Time Frame: Baseline and 12 months
Population: The analysis included all randomized participants who were included in the primary analysis aside from n=1 control who did not attend MRI appointment at 12-months.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Number analyzed (Participants) | 4 | 9
ratio
  NAA Baseline | 3.76 (0.16) | 3.96 (0.11)
  NAA 12 Months | 3.87 (0.16) | 3.89 (0.11)
  Cr Baseline | 3.09 (0.16) | 2.91 (0.11)
  Cr 12 Months | 3.24 (0.16) | 3.08 (0.11)
  Cho Baseline | 1.42 (0.14) | 1.45 (0.09)
  Cho 12 Months | 1.59 (0.14) | 1.55 (0.09)
  mIo Baseline | 1.10 (0.22) | 1.19 (0.15)
  mIo 12 Months | 0.88 (0.22) | 1.07 (0.15)
Statistical Analysis 1: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in NAA/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.49, ANOVA
Statistical Analysis 2: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in Cr/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.94, ANOVA
Statistical Analysis 3: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in Cho/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.80, ANOVA
Statistical Analysis 4: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in mIo/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.72, ANOVA

4. Secondary Outcome: Change in MRS Cerebral Metabolite Ratios in Frontal White Matter
Description: Change in major cerebral metabolites in the frontal white matter, as measured by 1H-Magnetic Resonance Spectroscopy (MRS), between baseline and 12-months. Spectra were acquired on a Phillips Achieva 3T MRI scanner using point-resolved spectroscopy (PRESS) sequence with short TE. jMRUI/AMARES algorithm was used to process spectra. Metabolite ratios were calculated for the following metabolites: N-acetyl aspartate (NAA), choline (Cho), creatine (Cr), myo-inositol (mIo), glutamate/glutamine complex (Glx), in relation to internal H2O as standard.
Time Frame: Baseline and 12 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Number analyzed (Participants) | 4 | 9
ratio
  NAA Baseline | 4.32 (0.34) | 4.16 (0.23)
  NAA 12 Months | 4.30 (0.34) | 4.16 (0.23)
  Cr Baseline | 2.74 (0.21) | 2.93 (0.14)
  Cr 12 Months | 2.99 (0.21) | 3.05 (0.14)
  Cho Baseline | 2.19 (0.16) | 2.13 (0.11)
  Cho 12 Months | 2.19 (0.16) | 2.24 (0.11)
  mIo Baseline | 1.11 (0.15) | 1.07 (0.10)
  mIo 12 Months | 1.15 (0.15) | 1.35 (0.10)
  Glx Baseline | 2.16 (0.23) | 2.27 (0.15)
  Glx 12 Months | 2.05 (0.23) | 2.18 (0.15)
Statistical Analysis 1: Comparison: Standard of Care HAART Regimen vs Maraviroc; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.95, ANOVA
Statistical Analysis 2: Comparison: Standard of Care HAART Regimen vs Maraviroc; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.66, ANOVA
Statistical Analysis 3: Comparison: Standard of Care HAART Regimen vs Maraviroc; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.56, ANOVA
Statistical Analysis 4: Comparison: Standard of Care HAART Regimen vs Maraviroc; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.29, ANOVA
Statistical Analysis 5: Comparison: Standard of Care HAART Regimen vs Maraviroc; Change in Glx/H20 levels were analysed using repeated-measures ANOVA with arm, time, and arm*time interaction as fixed effects; Test type: Superiority or Other; p = 0.95, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline to 12-months
Arm/Group | Standard of Care HAART Regimen | Maraviroc
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 2/8 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care HAART Regimen (N=8) | Maraviroc (N=9)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Small pilot sample size (N=17).
2. Unrepresentative of international HAND populations.
3. Open-label design may have contributed to loss to follow-up in controls.
4. Modified intention-to-treat design potentially introduced bias into analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less